CLINICAL TRIAL: NCT07159984
Title: The Effect of Training Given to Pregnant Women and Their Partners on Coping With Stress as a Couple, Couple Adjustment, Complaints and Quality of Life: A Randomized Controlled Study
Brief Title: Training Given to Pregnant Women and Their Partners on Coping With Stress as a Couple, Couple Adjustment, Complaints and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Burcu KUCUKKAYA, Assoc. Prof., Trakya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025-SBB-0331
Record Dates: First submitted 2025-08-30; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Pregnant Women; Coping With Stress as a Couple; Dyadic Adjustment; Complaints; Quality of Life; Education; Pregnancy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education group (Experimental)
  Interventions: Behavioral: Education on Changes During Pregnancy
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Education on Changes During Pregnancy — In the first session of the researcher-prepared training presentation, women will be informed about the structure and functions of their internal and external reproductive organs, as well as changes in physical, hormonal, social, and lifestyle activities. After the first session, there will be a 15-minute break before the second session, which will include evidence-based training on the effects of pregnancy-related changes on stress, couple harmony, and quality of life. Methods for coping with stress and pregnancy-related complaints, process management that positively impacts couple harmony, and healthy lifestyle behaviors that enhance quality of life will be discussed.
  Arms: Education group

SUMMARY:
Objective: This study aims to examine the effect of education provided to pregnant women and their partners on coping with stress as a couple, couple harmony, complaints, and quality of life regarding changes during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women and their spouses who are over 18 years of age,
* Literate and able to understand Turkish,
* Married,
* With a living spouse,
* Primiparous,
* Who have applied to the Bartın Provincial Health Directorate Healthy Life Center Pregnancy Class,
* Have written consent, and volunteer to participate in the study

Exclusion Criteria:

* Those who withdrew or dropped out of the study early,
* Those who were not willing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2025-05-18 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
The Couple Coping Inventory | change from Baseline (before implementation) and at 1st and 4th weeks of practice
  Developed by Bodenmann to measure couple coping and stress communication in romantic relationships . The inventory is a 5-point Likert-type scale with 37 items. Item scores range from 1 (never) to 5 (always).
The Pregnancy Complaints and Their Impact on Quality of Life Scale | change from Baseline (before implementation) and at 1st and 4th weeks of practice
  This scale measures pregnancy complaints and their impact on quality of life. The scale contains 42 items and consists of two sections. The first section assesses the frequency of pregnancy-related complaints experienced in the past month, and the second section assesses how these complaints impact daily activities. As the total score increases, quality of life decreases.
The Revised Dyadic Adjustment Scale | change from Baseline (before implementation) and at 1st and 4th weeks of practice
  The RDS is the final version of the 32-item Dyadic Adjustment Scale developed by Spanier, which was revised and reduced to 14 items.

CONTACTS AND LOCATIONS:
Locations (1):
- Eskişehir Osmangazi University, Eskişehir, Turkey (Türkiye)